CLINICAL TRIAL: NCT03464227
Title: A Subject-Blind, Investigator-Blind, Randomized, Placebo-Controlled, First-in-Human Study to Evaluate Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous Doses of UCB0107 in Healthy Male Subjects
Brief Title: A Study to Test the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous Doses of UCB0107 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0047; 2017-003315-19 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-03-13 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy Male Volunteers
Keywords: Phase 1; UCB0107

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCB0107 (Experimental): Subjects randomized to this arm will receive UCB0107. This arm will consist of a maximum of 7 cohorts. The dose for cohort 1 will be fixed, proposed doses for cohorts 2,3,4,5,6 and 7 may be adapted based upon recommendation by the Safety Review Group.
  Interventions: Drug: UCB0107
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive matching Placebo to UCB0107. This arm will consist of a maximum of 7 cohorts.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB0107 — * Pharmaceutical form: solution for infusion
  * Route of administration: intravenous use
  Arms: UCB0107
Other: Placebo — * Pharmaceutical form: intravenous infusion
  * Route of administration: intravenous use
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending doses of UCB0107 administered by intravenous (iv) infusion in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male, >= 18 and <= 75 years of age
* Subject has a body mass index (BMI) >= 18.0 and < 30.0 kg/m^2, with a body weight of at least 50 kg and maximum 100 kg
* Subject is in good physical and mental health
* Subject has clinical laboratory test results within the reference ranges of the laboratory
* Subject's electrocardiogram (ECG) is considered "normal," or "abnormal" but clinically non-significant (as interpreted by the investigator)
* Male subject confirms that, during the study period and for a period of 6 months or 5 half-lives of the investigational medicinal product (IMP) (whichever is longer), when having sexual intercourse with a woman of childbearing potential, a method of efficient contraception will be used, including a barrier AND an additional highly effective contraceptive method by the female partner

Exclusion Criteria:

* Subject is an employee or direct relative of an employee of the contract research organization (CRO) or UCB
* Subject has previously been assigned to treatment in this study or in another study of the medication under investigation in this study
* Subject is considered to be a vulnerable participant
* Subject has had major surgery (including joint surgery) within 6 months prior to Screening, or has planned surgery within 6 months after study treatment
* Subject has an active infection (eg, sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 4 weeks before the first dose of IMP

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The incidence of Adverse Events (AEs) during the study | During the study from Visit 1 up to the Safety Follow-Up Visit (Week 20)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

SECONDARY OUTCOMES:
The Maximum concentration (Cmax) for UCB0107 in serum and cerebrospinal fluid | Pharmacokinetic samples and samples from cerebrospinal fluid will be taken at pre-defined time points throughout study completion (up to Week 20)
  Cmax: maximum observed serum concentration
The area under the concentration-time curve from time 0 to infinity (AUC) in serum and cerebrospinal fluid | Pharmacokinetic samples and samples from cerebrospinal fluid will be taken at pre-defined time points throughout study completion (up to Week 20)
  AUC: area under the concentration-time curve from time 0 to infinity
The area under the concentration-time curve from time 0 to time t, the time of the last quantifiable concentration (AUC(0-t)) in serum and cerebrospinal fluid | Pharmacokinetic samples and samples from cerebrospinal fluid will be taken at pre-defined time points throughout study completion (up to Week 20)
  AUC(0-t): area under the concentration-time curve from time 0 to time t, the time of the last quantifiable concentration
The time to maximum concentration (tmax) for UCB0107 in serum and cerebrospinal fluid | Pharmacokinetic samples and samples from cerebrospinal fluid will be taken at pre-defined time points throughout study completion (up to Week 20)
  tmax: time to maximum observed serum concentration
The terminal half-life (t½) of UCB0107 in serum | Pharmacokinetic samples will be taken at pre-defined time points throughout study completion (up to Week 20)
  t1/2: terminal half-life
The total Clearance (CL) for UCB0107 in serum | Pharmacokinetic samples will be taken at pre-defined time points throughout study completion (up to Week 20)
  CL: clearance
The volume of distribution (Vz) for UCB0107 in serum | Pharmacokinetic samples will be taken at pre-defined time points throughout study completion (up to Week 20)
  Vz: volume of distribution.
CSF/serum ratio of antibody concentrations | Pharmacokinetic samples and samples from cerebrospinal fluid will be taken at pre-defined time points throughout study completion (up to Week 20)
  Ratio of the antibody concentrations in cerebrospinal fluid and serum

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0047 001, Berlin, Germany